CLINICAL TRIAL: NCT03592966
Title: Randomised, Double-blind, Placebo Controlled, Crossover Trial Investigating the Acute Effects of Blueberry (Poly)Phenols on Vascular Function and Cognitive Performance in Healthy Individuals Across the Life Course.
Brief Title: Investigating the Acute Effects of Blueberry (Poly)Phenols on Vascular Function and Cognition in Healthy Individuals.
Acronym: BluLife
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Reading (Other)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Principal Investigator, King's College London
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: BLULIFE
Record Dates: First submitted 2018-04-06; First posted 2018-07-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-05

CONDITIONS: Healthy
Keywords: (Poly)phenols; Blueberries; Anthocyanins; Cognitive function; Vascular function

STUDY DESIGN:
Intervention Model Description: Randomized, cross-over, double-blind, placebo-controlled study.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Freeze-dried placebo powder
  Interventions: Dietary Supplement: Placebo
- Wild Blueberry powder (Active Comparator): Freeze-dried whole fruit blueberry drink.
  Interventions: Dietary Supplement: Wild Blueberry Powder

INTERVENTIONS:
Dietary Supplement: Wild Blueberry Powder — Freeze-dried whole fruit blueberry drink.
  Arms: Wild Blueberry powder
Dietary Supplement: Placebo — Freeze-dried placebo powder
  Arms: Placebo

SUMMARY:
This study aims to determine the effect of blueberry (poly)phenol vs placebo on vascular function and cognitive performance with an insight into cerebral blood flow velocity changes, across all ages of the general healthy population.

DETAILED DESCRIPTION:
Foods rich in certain (poly)phenols, particularly flavonoids, such as berries, have been shown to improve measures of vascular function as well as cognitive performance in human intervention studies. Blueberries are rich in anthocyanins, a subclass of flavonoids that have been widely linked to health benefits, particularly improvements in endothelial function. Research have previously shown that blueberries improve executive functioning and memory in both healthy adults and children. These improvements were seen within 2-5 hours post-consumption of blueberries, a time-course that positively correlates with improvements in vascular function (measured as flow-mediated dilation). This indicates that increases in blood flow may influence improvements in cognitive performance. To date no study has investigated whether blueberry consumption can induce an increase in cerebral blood flow, with subsequent improvements in vascular and cognitive function. In this study, investigators aim to directly link wild blueberry consumption with increased vascular and cerebral blood flow and positive cognitive outcomes in healthy individuals through the life course, between the ages of 8 and 80 years old. Investigators will use a large group of healthy subjects representative of the general public over a wide age range in males and females to evaluate the generalisability of the health benefits of blueberry consumption.

ELIGIBILITY:
Inclusion criteria:

* Healthy men and women aged 8-80 years old
* Are able to understand the nature of the study
* Able and willing to give signed written informed consent with the addition of a parent/carer for the consent of children under 16.
* Are willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study.

Exclusion Criteria:

* Manifest cardiovascular diseases including coronary artery disease, cerebrovascular disease and peripheral artery disease.
* Hypertensive, as defined as SBP superior or equal to 140 mmHg or DBP superior or equal to 90 mmHg.
* Obese participants, defined as BMI superior or equal to 30.
* Diabetes mellitus and metabolic syndrome.
* Acute inflammation, terminal renal failure or malignancies.
* Abnormal heart rhythm (lower or higher than 60-100 bpm).
* Allergies to berries or another significant food allergy.
* Subjects under medication or on vitamin/dietary supplements (within 2 weeks of baseline).
* Subjects who have lost more than 10% of their weight in the past 6 months or are currently on a diet.
* Subjects who reported participant in another study within one month before the study starts.
* Subjects who smoke cigarettes.
* MCI or dyslexic or unable to complete the cognitive function tasks for any reason such as visual impairments.
* Subjects who require chronic antimicrobial or antiviral treatment.
* Subjects with unstable psychological condition.
* Subjects with history of cancer, myocardial infarction, cerebrovascular incident.
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Cognitive function | Change from baseline cognitive function at 2 hours post-consumption
  Cognitive testing involves the participant conducting tasks administered on a tablet-style laptop. The participants will be conducting these tasks whilst cerebral blood flow measurements are taking place. The cognitive testing battery will consist of 4 tasks including a mood assessment (PANAS).
Endothelial Function | Change from baseline endothelial function at 2 hours post-consumption
  Flow mediated dilation (FMD)

SECONDARY OUTCOMES:
Cerebral blood flow (CBF) | Change of baseline cerebral blood flow at 2 hours post consumption
  Trans-cranial blood flow will be assessed by Non-imaging transcranial Doppler sonography (TCD)
Blood pressure | Change from baseline systolic blood pressure at 2 hours post consumption
  Automated clinical digital sphygmomanometer

OTHER OUTCOMES:
Plasma blueberry (poly)phenol metabolites | 2 hours
  Measured by liquid chromotography- mass spectrometry (LC/MS)
Urine (poly)phenol metabolites | Baseline and 12 weeks
  24-hour urine samples

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom